CLINICAL TRIAL: NCT03846531
Title: Evaluation of Nano-Pulse Stimulation (NPS) in Patients With Seborrheic Keratosis
Brief Title: Nano-Pulse Stimulation (NPS) in Seborrheic Keratosis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NP-SK-002
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Lesion Skin; Seborrheic Keratosis
Keywords: Nano-Pulse Stimulation; Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Intervention Model Description: Each subject served as their own control. Each subject had 4 lesions with 3 of the lesions serving in the Active Comparative Arm (Lesions treated with Nano-Pulse Stimulation) and 1 lesion serving as control not treated with Nano-Pulse Stimulation and assigned to No Intervention Arm.
Who Masked: Outcomes Assessor
Masking Description: A Reference Key was developed for 3 independent reviewers to use during their review of the full set (196 image pairs) of study photographs. The reference key included 2 representative photographs for each of the 4 possible scores used in the SK study (clear, mostly clear, partially clear, and not clear). The three independent reviewers were not principal investigators at enrolling centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Nano-Pulse Stimulation (NPS) Lesion (Active Comparator): Three of four selected SK lesions receive Nano-Pulse Stimulation treatment.
  Interventions: Device: Nano-Pulse Stimulation (NPS)
- Non-Treated Lesion (No Intervention): One of four SK lesions is randomized to not receiving Nano-Pulse Stimulation treatment.

INTERVENTIONS:
Device: Nano-Pulse Stimulation (NPS) — The Pulse generator delivers electrical pulses (nanosecond duration) that are applied directly to targeted lesion using sterile treatment tips with micro-needles.
  Arms: Nano-Pulse Stimulation (NPS) Lesion

SUMMARY:
The primary purpose of this trial is to evaluate Nano-Pulse Stimulation (NPS) to clear or remove Seborrheic Keratosis (SK) lesions from off-facial areas of healthy adult subjects.

DETAILED DESCRIPTION:
Evaluate Nano-Pulse Stimulation (NPS) to clear or remove Seborrheic Keratosis (SK) lesions from off-facial areas of healthy adult subjects.

The specific objectives of this study are to:

* Document the non-treated appearance of off-face SKs.
* Evaluate the clearance of SKs in off-face locations post-treatment versus pre-treated appearance of the same lesion.
* Evaluate the clearance of the treated SKs at various points in time over several weeks following the initial procedure, compared to the pre-treated SKs.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent
* Has a clinical diagnosis of stable, clinically typical seborrheic keratosis
* Medically determined candidate for at least 4 off-face SK lesions
* Must have at least four treatable SK lesions and be willing to have NPS treatment on any three of the four treatable SK lesions. Treatable SK lesions must: be at least 1 mm in height, and no greater than 3 mm in height and not have a dimension perpendicular to the longest dimension of greater than 7.5mm or longer in any dimension than 20mm
* Willing to have three of the designated SK lesions treated in a single treatment session
* Willing to return to the PI's office for five additional study visits at specified intervals over 106-days
* Agrees to high resolution photos of both the treated SK lesions and the untreated SK lesion
* No subject identity will be possible via the "lesion-only" photograph
* No evidence of active infection in the designated tissue prior to treatment
* Is not allergic to Lidocaine or Lidocaine-like products
* Not pregnant or lactating

Exclusion Criteria:

* Has an implantable electronic device (e.g., automatic defibrillator)
* Active infection or history of infection within 90 previous days in designated test area
* Not willing or able to sign the Informed Consent
* Non-English speaking or reading
* Is known to be immune-compromised
* Known to be a keloid producer
* On blood thinning medications
* Diseases, conditions, or situations wherein the PI judges that the patient is not appropriate for participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (4):
- United States (4):
  - Premier Plastic Surgery, San Mateo, California
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - Zel Skin & Laser Specialists, Edina, Minnesota
  - Laser & Dermatologic Surgery Center, Chesterfield, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hruza GJ, Zelickson BD, Selim MM, Rohrer TE, Newman J, Park H, Jauregui L, Nuccitelli R, Knape WA, Ebbers E, Uecker D. Safety and Efficacy of Nanosecond Pulsed Electric Field Treatment of Seborrheic Keratoses. Dermatol Surg. 2020 Sep;46(9):1183-1189. doi: 10.1097/DSS.0000000000002278. PMID 31809349

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4 SK study lesions were enrolled per subject, one SK lesion was randomized to be an internal subject control and the 3 other SK lesions were pre-assigned for treatment for a total of 232 study lesions; 58 Controls and 174 Treated lesions.
Units Other Than Participants: SK lesions
Groups:
- Nano-Pulse Stimulation (NPS) Treatment Arm: Three of four selected SK lesions receive Nano-Pulse Stimulation treatment.
  Nano-Pulse Stimulation (NPS): The Pulse generator delivers electrical pulses (nanosecond duration) that are applied directly to targeted lesion using sterile treatment tips with micro-needles.
Period: Overall Study
Arm/Group | Nano-Pulse Stimulation (NPS) Treatment Arm
Started | 58; 174 SK lesions
Completed | 58; 174 SK lesions
Not Completed | 0; 0 SK lesions

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes 58 Participants with 3 treated SK lesions and one SK lesion as an internal control for a total of 4 SK lesions per participants.
Units Other Than Participants: SK lesions
Arm/Group | Nano-Pulse Stimulation (NPS) Lesion
Number analyzed (Participants) | 58
Number analyzed (SK lesions) | 174
Age, Continuous [Mean (Full Range); unit: years] | 61 [34 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Clearance of SK Lesions
Description: Total Number of treated SK lesions per participant rated as clear or mostly-clear by the Principal Investigator at each clinical site.
Time Frame: 106-day post-treatment
Population: Fifty-eight (58) participants with each participant having a total of 4 SK lesions, 3 treated and 1 serving as an internal untreated control.
Measure: Number; unit: percentage of SK lesion clearance
Units Other Than Participants: SK lesions
Arm/Group | Nano-Pulse Stimulation (NPS) Lesion
Number analyzed (Participants) | 58
Number analyzed (SK lesions) | 174
percentage of SK lesion clearance | 82

ADVERSE EVENTS:
Time Frame: 3.5 months (106 days)
Groups:
- Nano-Pulse Stimulation (NPS) Treatment Arm: Three of four selected SK lesions received Nano-Pulse Stimulation treatment.
  Nano-Pulse Stimulation (NPS): The Pulse generator delivers electrical pulses (nanosecond duration) that are applied directly to targeted lesion using sterile treatment tips with micro-needles.
Arm/Group | Nano-Pulse Stimulation (NPS) Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 35/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nano-Pulse Stimulation (NPS) Treatment Arm (N=58)
Transient Hyperpigmentation (Skin and subcutaneous tissue disorders) | 35 (35) — Skin hyperpigmentation at the site of treated lesion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT03846531/Prot_SAP_001.pdf